CLINICAL TRIAL: NCT01036074
Title: Reward Processing in Cocaine Addiction
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905399; 05-DA-N399
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-04-08

CONDITIONS: Drug Abuse; Cocaine Dependence
Keywords: Drug Abuse; Cocaine; Cocaine Dependence; Functional MRI; Pharmalogical MRI; Conditioning
MeSH Terms: conditions — Substance-Related Disorders; Cocaine-Related Disorders

SUMMARY:
Background:

- Cocaine affects the brain's ability to process information. However, different people respond to cocaine in different ways, and differences in brain structure and function may affect how cocaine alters brain activity. By using functional magnetic resonance imaging (fMRI) to monitor brain activity during tasks that provide simple rewards, researchers hope to better understand how the brain responds to rewards and how this response is affected by drugs like cocaine.

Objectives:

* To determine the effect of cocaine administration on the reward experience in cocaine-dependent individuals.
* To study genetic and personality factors that may contribute to cocaine dependence.

Eligibility:

- Individuals between 18 and 45 years of age who either are cocaine-dependent and not seeking treatment or are healthy volunteers.

Design:

* Participants will be asked to avoid consuming alcohol and restrict consumption of caffeine prior to the study. Participants provide urine and breath samples to be tested for chemicals that may interfere with the study.
* All participants will complete a training session and at least one fMRI scanning session. During the training session, participants will be introduced to the reward tasks and MRI equipment.
* Healthy volunteers will have a single fMRI session that will involve reward tasks to be completed during the scanning. Rewards will include small amounts of fruit juice and the opportunity to win money.
* Cocaine-dependent participants will have a training session and three experimental sessions including 1) a mock MRI scan to test cocaine tolerance, 2) one fMRI scan with reward tasks after administration of IV cocaine, and 3) one fMRI scan with reward tasks after administration of IV placebo (saline solution). Rewards will include small amounts of fruit juice and the opportunity to win money.
* In addition to the scans, participants will provide a blood sample for further study and will answer questionnaires provided by the researchers.

DETAILED DESCRIPTION:
Objective:

The overall objective of this study is to determine the effect that cocaine administration has upon the experience of reward in dependent individuals and the contribution of reward processing (or dysfunction) to the reinforcing effects of cocaine and the recidivism rates noted in cocaine-dependent individuals. The primary goal is to employ functional magnetic resonance imaging (fMRI) to ascertain the function of neural systems that respond to cocaine in human participants and to determine the role that they play in the processing of different types of rewarding stimuli during episodes where individuals are drug-free and those where they are under the acute influence of cocaine.

Study Population:

The experimental population for this investigation will be non-treatment seeking, cocaine-dependent adults (i.e. 18 45 years old). A cohort of healthy, drug-free, individuals, matched for age, gender, ethnicity and IQ, will serve as a control group.

Design:

This experiment employs a mixed-measures, counter-balanced design. Participants will complete two measures of reward processing (i.e. the revised monetary incentive delay (MID) task and a temporal difference error task (TDE/juice) task) while undergoing BOLD EPI fMRI. The scanning procedure will be repeated for all subjects, such that each participant undertakes 2 sessions. Cocaine-dependent individuals will receive either two injections of cocaine (30 mg/70 kg body weight; intravenous (IV) administration) or two injections of saline during scanning. Within each session, each IV injection will be given approximately 10 minute prior to the start of one of the reward measures. The order of cocaine and saline scans will be randomized and participants will be blind to the experimental condition prior to participation.

Outcome Measures:

The primary outcome measures will be the neural substrates of reward processing and how these differ between cocaine-dependent individuals and controls, and the impact of acute cocaine administration upon brain function associated with reward function.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALL PARTICIPANTS

Participants in both groups must be:

1. Generally healthy.
2. Right handed.
3. Males or non-pregnant/non-lactating females.
4. Between the ages of 18-45, for cocaine dependent participants; 18-50 for control participants.

Cocaine-dependent participants must also:

1. Meet DSM-IV criteria for dependence at the time of participation.
2. Be positive for cocaine use in their urine toxicology screen either at their screening visit or on another occasion prior to their entry to the study (please note that this could be as late as the day of study entry).
3. Use either injection or smoking as their primary route of cocaine administration.

EXCLUSION CRITERIA:

ALL PARTICIPANTS

Participants in both groups will be excluded from participation in this study if they:

1. Are unable to undergo MRI scanning due to pregnancy, implanted metallic devices (e.g. cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; or other implanted metal parts), or claustrophobia.
2. Suffer from any major medical illness that may effect central nervous function including (but not limited to): hypertension; clinically significant arrhythmia; cardiovascular disease; asthma; diabetes; peripheral vascular diseases; coagulopathies; history of superficial or deep vein thrombosis; HIV; or syphilis.
3. Have any neurological illnesses including (but not limited to): seizure disorders; migraine; multiple sclerosis; movement disorders; or history of head trauma, CVA, or CNS tumor.
4. Have a history of syncope
5. Have an estimated IQ of < 85
6. Are lactating or pregnant
7. Are currently taking any psychoactive or vasoactive medication(s).
8. Meet DSM-IV criteria for dependence on alcohol or marijuana. Recreational use of alcohol and/or marijuana will be tolerated in all participants as will nicotine dependence.

COCAINE-DEPENDENT PARTICIPANTS

Cocaine-dependent individuals will also be excluded from participation if:

They have any current or previous history of any major psychiatric disorder other than cocaine dependence, including but not limited to mood, anxiety and psychotic disorders.

They have current dependence on any substance of abuse, other than cocaine or nicotine. However, current or past co-morbid abuse of alcohol, marijuana and past dependence on other substances of abuse will be tolerated in this group.

They have a history of adverse reaction to cocaine, such as cardiac arrhythmia or chest pain.

CONTROL PARTICIPANTS

Control participants will be excluded if they:

1. Are currently, or have previously been, dependent on alcohol or any other drug (with the exception of nicotine).
2. Meet the DSM-IV criteria for substance abuse of any substance.
3. Have any current, or previous, diagnosis of any major psychiatric disorder, i.e. to include (but not limited to) mood, anxiety, and psychiatric disorders, or any substance-induced psychiatric disorders.
4. Have any family history of psychosis (based on self-report).
5. Have previously been diagnosed with a DSM-IV Axis II disorder.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2005-03-17; Study Completion 2013-04-08

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Akil M, Kolachana BS, Rothmond DA, Hyde TM, Weinberger DR, Kleinman JE. Catechol-O-methyltransferase genotype and dopamine regulation in the human brain. J Neurosci. 2003 Mar 15;23(6):2008-13. doi: 10.1523/JNEUROSCI.23-06-02008.2003. PMID 12657658
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Balster RL, Schuster CR. Fixed-interval schedule of cocaine reinforcement: effect of dose and infusion duration. J Exp Anal Behav. 1973 Jul;20(1):119-29. doi: 10.1901/jeab.1973.20-119. PMID 4197505